CLINICAL TRIAL: NCT03576027
Title: Evaluation of the Effectiveness of Hyperbaric Oxygen Therapy in the Treatment of Inflammatory Bowel Disease in Children
Brief Title: Hyperbaric Oxygen Therapy in Children With Inflammatory Bowel Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Lukasz Dembinski, Principal Investigator, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dembinski2018
Record Dates: First submitted 2018-06-10; First posted 2018-07-03 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Inflammatory Bowel Diseases; Children, Only
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperbaric oxygen therapy (Experimental)
  Interventions: Other: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — Hyperbaric Oxygen Therapy

SUMMARY:
The study assesses the effectiveness of hyperbaric oxygen therapy in the treatment of inflammatory bowel disease in children.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Crohn's disease or ulcerative colitis according to the criteria from Porto - based on the clinical condition as well as imaging and endoscopic examinations with histopathological assessment;
* failure to achieve the remission despite the use of standard treatment in accordance with international guidelines;
* written consent of the patient's legal guardians and the patient himself if he/she turns 16 years of age.

Exclusion Criteria:

* intolerance of enclosed spaces;
* contraindications for hyperbaric therapy: otolaryngological (otitis media, sinusitis); cardiac (clinically significant defects or arrhythmias); pneumological (clinically significant defects)
* exacerbation of inflammatory bowel disease during the therapy;
* contraindications for hyperbaric therapy in a patient's caregiver in a situation, where the patient requires his/hers presence inside the hyperbaric chamber during the session.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the ulcerative colitis activity | 40 days
  Change in the disease activity based on the Paediatric Ulcerative Colitis Activity Index (PUCAI) for patients with ulcerative colitis.
Change of the Crohn's disease activity | 40 days
  Change in the disease activity based on the Pediatric Crohn's Disease Activity Index (PCDAI) for patients with Crohn's disease.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 40 days
  Number of participants with treatment-related adverse events and the the severity of these events.
Concentration of proinflammatory cytokines | 40 days
Maintaining remission of the ulcerative colitis | 1 year
  Duration of the clinical remission time (if achieved) assessed according to the Paediatric Ulcerative Colitis Activity Index (PUCAI) for patients with ulcerative colitis.
Maintaining remission of the Crohn's disease | 1 year
  Duration of the clinical remission time (if achieved) assessed according to the Pediatric Crohn's Disease Activity Index (PCDAI) for patients with Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Dembinski, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No